CLINICAL TRIAL: NCT06982469
Title: Magnetic Resonance Imaging (MRI)/ Positron Emission Tomography (PET) Prostate-specific Membrane Antigen (PSMA) -Based Phase I-II Study of Salvage HDR Brachytherapy and External Beam Irradiation In Isolated Tumor Bed Relapses After Radical Prostatectomy
Brief Title: High Dose Rate (HDR) Brachytherapy Salvage After Prostatectomy
Status: Recruiting | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: 2020.212
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer; Prostatectomy; Local Recurrence of Malignant Tumor of Prostate; Radiotherapy; Complications; Brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort 1: Patients with increasing prostatic specific antigen (PSA) after radical prostatectomy (RP) and clinical evidence of PET PSMA+ and MRI (magnetic resonance imaging)+ isolated prostatic bed relapse (IPBR) that is implantable via transperineal route . The IPBR should be visible on TRUS imaging to allow proper implant placement
  Interventions: Radiation: Brachytherapy

INTERVENTIONS:
Radiation: Brachytherapy — HDR brachytherapy

SUMMARY:
The goal of this observational study is to learn about the long-term effects of HDR Brachytherapy in men with isolated local relapses after radical prostatectomy. The main question it aims to answer is:

Does HDR Brachytherapy increase control rates and decreases complications compared with conventional External Irradiation?

Participants will be asked to receive HDR brachytherapy as part of their regular medical care for isolated local relapses after radical prostatectomy

DETAILED DESCRIPTION:
HDR brachytherapy appears to be an ideal technique for dose escalation in PET/MRI+ (positron emission tomography) , small, well-defined IPBR that can be accessed and visualized through the perineal route with transrectal ultrasound (TRUS) guidance. Additionally, HDR brachytherapy can spare from high dose irradiation most of the vesicourethral anastomosis, the external urinary sphincter (EUS) and the penile bulb. This may be crucial in circular structures such as EUS that are particularly sensitive to whole-volume irradiation but tolerate well high small-volume doses provided that the rest of the EUS is spared.

In this study, HDR brachytherapy will be combined with external beam radiation and 6 months of androgen deprivation therapy to decrease the prostate bed volume irradiated at high-doses while increasing the radiation dose in the PET/MRI+ areas.

ELIGIBILITY:
Inclusion Criteria:

* Patients with increasing PSA after RP and clinical evidence of PET PSMA/Choline+ and MRI+ isolated prostatic bed relapse (IPBR) that is implantable via transperineal route . The IPBR should be visible on TRUS imaging to allow proper implant placement.
* Pathological confirmation is advised in all cases but it is not mandatory .
* Brachytherapy MRI-based dosimetry
* Patient written Informed Consent of the Institutional Review Board-approved protocol that discloses the investigational nature of the treatment as well as the available standard treatment options.

Exclusion Criteria:

* Distant Metastases
* Isolated nodal relapses
* Prior Irradiation to the IPBR area
* Multicentric IPBRs
* Life expectancy of less than 5 years or inability to tolerate and comply with an HDR procedure

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with isolated tumor bed relapses after radical prostatectomy
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
biochemical relapse-free survival (bRFS) | 5-year
  Biochemical Relapse-Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Martínez-Monge, M.D., Principal Investigator — Clinica Universidad de Navarra Cancer Center
Locations (1):
- Clínica Universidad de Navarra, Pamplona, Foral Community of Navarre, Spain

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, ICF
Time Frame: After Primary Completion
Access Criteria: On request

REFERENCES:
- [Background] Carrie C, Magne N, Burban-Provost P, Sargos P, Latorzeff I, Lagrange JL, Supiot S, Belkacemi Y, Peiffert D, Allouache N, Dubray BM, Servagi-Vernat S, Suchaud JP, Crehange G, Guerif S, Brihoum M, Barbier N, Graff-Cailleaud P, Ruffion A, Dussart S, Ferlay C, Chabaud S. Short-term androgen deprivation therapy combined with radiotherapy as salvage treatment after radical prostatectomy for prostate cancer (GETUG-AFU 16): a 112-month follow-up of a phase 3, randomised trial. Lancet Oncol. 2019 Dec;20(12):1740-1749. doi: 10.1016/S1470-2045(19)30486-3. Epub 2019 Oct 16. PMID 31629656
- [Background] Gonzalez-San Segundo C, Counago F, Gomez-Iturriaga A. Androgen Deprivation Therapy and Salvage Radiotherapy: Are We Missing Something? Eur Urol. 2019 Aug;76(2):260-261. doi: 10.1016/j.eururo.2019.01.045. Epub 2019 Feb 8. No abstract available. PMID 30745145
- [Background] Carrie C, Hasbini A, de Laroche G, Richaud P, Guerif S, Latorzeff I, Supiot S, Bosset M, Lagrange JL, Beckendorf V, Lesaunier F, Dubray B, Wagner JP, N'Guyen TD, Suchaud JP, Crehange G, Barbier N, Habibian M, Ferlay C, Fourneret P, Ruffion A, Dussart S. Salvage radiotherapy with or without short-term hormone therapy for rising prostate-specific antigen concentration after radical prostatectomy (GETUG-AFU 16): a randomised, multicentre, open-label phase 3 trial. Lancet Oncol. 2016 Jun;17(6):747-756. doi: 10.1016/S1470-2045(16)00111-X. Epub 2016 May 6. PMID 27160475
- [Background] Martinez-Monge R, Moreno M, Ciervide R, Cambeiro M, Perez-Gracia JL, Gil-Bazo I, Gaztanaga M, Arbea L, Pascual I, Aristu J. External-beam radiation therapy and high-dose rate brachytherapy combined with long-term androgen deprivation therapy in high and very high prostate cancer: preliminary data on clinical outcome. Int J Radiat Oncol Biol Phys. 2012 Mar 1;82(3):e469-76. doi: 10.1016/j.ijrobp.2011.08.002. PMID 22284039